CLINICAL TRIAL: NCT00767819
Title: Multicenter, Triple-arm, Single-stage, Phase II Trial to Determine the Preliminary Efficacy and Safety of RAD001 in Patients With Histological Evidence of Progressive or Metastatic Bone or Soft Tissue Sarcomas
Brief Title: Treatment of Patients With RAD001 With Progressive Sarcoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CRAD001C24114; 2007-005294-60 (EudraCT Number)
Record Dates: First submitted 2008-10-06; First posted 2008-10-07 (Estimated); Results first posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2018-12

CONDITIONS: Progressive Sarcoma
Keywords: progressive GIST; progressive sarcoma
MeSH Terms: interventions — Everolimus

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm 1 (Experimental): Progressive or metastatic bone or soft tissue sarcomas
  Interventions: Drug: Everolimus
- Arm 2 (Experimental): Progressive gastrointestinal stromal tumors (GIST) after failure of prior imatinib and sunitinib 1st and 2nd line
  Interventions: Drug: Everolimus
- Arm 3 (Experimental): Progressive or metastatic alveolar soft part sarcoma (ASPS)
  Interventions: Drug: Everolimus

INTERVENTIONS:
Drug: Everolimus — 2.5 and 5 mg tablets taken orally and starting dose was 10 mg daily for all patients
  Other Names: RAD001

SUMMARY:
The purpose of this multicenter, three-arm, exact binomial single-stage, phase II trial is to determine the preliminary efficacy and safety of RAD001 in patients with histological evidence of progressive or metastatic bone or soft tissue sarcoma.

ELIGIBILITY:
Inclusion Criteria:

Histological evidence of progressive or metastatic bone or soft tissue sarcoma.

The following tumor types are included:

* malignant fibrous histiocytoma
* liposarcoma
* synovial sarcoma
* malignant paraganglioma
* fibrosarcoma
* leiomyosarcoma
* angiosarcoma including haemangiopericytoma
* malignant peripheral nerve sheath tumor
* STS, not otherwise specified
* miscellaneous sarcoma including mixed mesodermal tumors of the uterus
* osteosarcoma
* Ewing's sarcoma
* rhabdomyosarcoma
* gastrointestinal stromal tumor (only after failure or intolerance of imatinib or sunitinib in 1st and 2nd line)
* alveolar soft part sarcoma (ASPS)

  * Objective progression of disease may be documented by RECIST criteria. Any of the following would be sufficient according to RECIST:
* a 20% increase in the sum of unidimensionally measured target lesions
* a new lesion
* unequivocal increase in non-measurable disease.

  * Patients must have disease not amenable to surgery, radiation, or combined modality therapy with curative intent.
  * ECOG performance status 0 - 2.

Exclusion Criteria:

Anticancer therapy within 3 weeks of enrollment including chemotherapy, hormonal therapy, immunotherapy, or radiotherapy.

* The following tumor types will not be included:

  * gastrointestinal stromal tumor (except for patients after treatment with imatinib or sunitinib in 1st and 2nd line)
  * chondrosarcoma
  * malignant mesothelioma
  * neuroblastoma.
* Prior therapy with RAD001 (everolimus) or other rapamycins (sirolimus, temsirolimus).
* Neurotoxicity > grade 2 CTC.
* Radiation of the lung.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-03-31 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (6):
- Germany (5):
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Düsseldorf
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Mannheim
  - Novartis Investigative Site, München
- Novartis Investigative Site, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Seventy-four patients were screened and seventy-one enrolled.
Period: Overall Study
Arm/Group | Arm 1 | Arm 2 | Arm 3
Started | 37 | 24 | 10
Intent to Treat (ITT) Analysis Set | 37 | 24 | 10
Safety Analysis Set (SAF) | 37 | 24 | 10
Completed | 12 | 5 | 10
Not Completed | 25 | 19 | 0
Not completed — Unsatisfactory therapeutic effect | 18 | 14 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Administrative problems | 0 | 1 | 0
Not completed — Death | 2 | 3 | 0
Not completed — Adverse Event | 2 | 0 | 0
Not completed — Abnormal lab values | 1 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1 | Arm 2 | Arm 3 | Total
Number analyzed (Participants) | 37 | 24 | 10 | 71
Age, Customized [Count of Participants; unit: Participants]
  < 65 years | 31 | 14 | 9 | 54
  >= 65 years | 6 | 10 | 1 | 17
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 6 | 31
  Male | 23 | 13 | 4 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 36 | 24 | 10 | 70
  Black | 1 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Best Overall Response Rates by Week 16 (ITT)
Description: The best overall response is the best response recorded from treatment start until disease progression/recurrence (both measurement and confirmation criteria). Best lesion response was defined by (Resist Criteria V1 for target and non-target lesions): Complete Response (CR)=at least two determinations of CR 4 weeks apart before progression, Partial Response (PR)=at least two determinations of CR 4 weeks apart before progression (and not qualifying for a CR), Stable Disease (SD)=at least one SD assessment >6 weeks after start of treatment and Progressive Disease (PD)=Progression or death due to underlying cancer ≤16 weeks after start of treatment. PD without radiologic evidence were classified as progression only, when clear evidence of clinical deterioration was available and patient discontinued due to "disease progression". Unknown (UNK) = all other cases.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 37 | 24 | 10
percentage of participants
  Complete Response | 0 | 0 | 0
  Partial Response | 0 | 0 | 0
  Stable Disease | 40.5 | 33.3 | 100.0
  Progressive Disease | 51.4 | 62.5 | 0
  Unknown | 8.1 | 4.2 | 0
Statistical Analysis 1: Comparison: Arm 1 vs Arm 2 vs Arm 3; Test type: Superiority — The lower limit of the confidence interval was used to support the decision in favor of p0 or p1: if the lower limit of the confidence interval overlapped p0, the hypothesis that p is greater than or equal to p1 could be rejected; on the other side, if the lower limit of the confidence interval excluded p0, the hypothesis that p is greater than or equal to p1 could be accepted; p = 0.1, Clopper-Person confidence interval; percentage of participants = 40.5, 80% CI 2-sided [29.5 to 52.4]

2. Secondary Outcome: Objective Tumor Response Rates (Complete Response and Partial Response) at Week 16 (ITT)
Description: The best overall response is the best response recorded from the start of the treatment until disease progression/recurrence (taking as reference for PD the smallest measurements recorded since the treatment started). In general, the patient's best response assignment will depend on the achievement of both measurement and confirmation criteria. Best lesion response was defined by (Resist Criteria V1 for target and non-target lesions).
Time Frame: Baseline up to approximately 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 37 | 24 | 10
percentage of participants
  Complete response | 0 | 0 | 0
  Partial response | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants With Duration of Response (CR, PR, SD) at 16 Weeks.
Description: Duration of response (CR, PR or SD) applied only to those patients whose best overall response was CR, PR or SD based on local radiologic assessments and was defined as the time from start of treatment to progression or death from underlying disease. Patients not experiencing progression or death at 16 weeks were censored with the date of their last tumor assessment. Duration of response was explored using the Kaplan-Meier method.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 15 | 8 | 10
percentage of participants | 60 | 62.5 | 100

4. Secondary Outcome: Percentage of Participants With Progression-free Survival (PFS) at 16 Weeks
Description: Progression-free Survival (PFS) was defined as the time from the date of start of treatment to the date of event defined as the first documented progression or death from any cause. If a patient had not had an event, PFS was censored at the date of the last adequate tumor assessment at week 16
Time Frame: 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 37 | 24 | 10
percentage of participants | 35.1 | 30.5 | 100.0

5. Secondary Outcome: Time to Progression (TTP) (ITT)
Description: Time to progression (TTP) was defined as the time from the date of start of treatment to the date of event defined as the first documented progression or death from underlying disease. If a patient had not had an event, TTP was censored at the date of the last adequate tumor assessment, which was the date of Visit 6 (Week 16) for the core phase and the last available tumor assessment for the follow-up phase. TTP was explored by using the Kaplan-Meier method.
Time Frame: Baseline up to 16 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 37 | 24 | 10
days | 57 [55 to 114] | 57 [32 to 135] | 499 [231 to 704]

6. Secondary Outcome: Percentage of Participants With Overall Survival (OS) at Week 16 (ITT)
Description: Overall survival (OS) was defined as the time from the date of start of treatment to death from any cause. If a patient was not known to have died (was alive), OS was censored at the date of the last contact, which was the date of Visit 6 (Week 16) for the core phase and the last available visit for the follow-up phase. OS was explored by using the Kaplan-Meier method. One death occurred in Arm 3 after Week 16.
Time Frame: Baseline up to 16 weeks
Measure: Number; unit: percentage of participants
Arm/Group | Arm 1 | Arm 2 | Arm 3
Number analyzed (Participants) | 37 | 24 | 10
percentage of participants | 68.8 | 56.9 | 100.0

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit) up to approximately 16 weeks
Groups:
- Arm I: Progressive or metastatic bone or soft tissue sarcomas
- Arm II: Progressive gastrointestinal stromal tumors (GIST) after failure of prior imatinib and sunitinib 1st and 2nd line
- Arm III: Progressive or metastatic alveolar soft part sarcoma (ASPS)
Arm/Group | Arm I | Arm II | Arm III
All-Cause Mortality (participants affected / at risk) | 8/37 | 4/24 | 1/10
Serious Adverse Events (participants affected / at risk) | 15/37 | 14/24 | 8/10
Other Adverse Events (participants affected / at risk) | 35/37 | 21/24 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=37) | Arm II (N=24) | Arm III (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 1 | 0 | 0
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 | 1 | 0
PANCYTOPENIA (Blood and lymphatic system disorders) | 1 | 0 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1 | 0
PERICARDIAL EFFUSION (Cardiac disorders) | 1 | 0 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 | 3 | 0
COLITIS (Gastrointestinal disorders) | 0 | 0 | 1
DIARRHOEA (Gastrointestinal disorders) | 1 | 0 | 0
NAUSEA (Gastrointestinal disorders) | 1 | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 0 | 1 | 0
VOMITING (Gastrointestinal disorders) | 1 | 3 | 0
ASTHENIA (General disorders) | 1 | 0 | 0
CHEST PAIN (General disorders) | 0 | 0 | 1
DISEASE PROGRESSION (General disorders) | 0 | 1 | 0
FATIGUE (General disorders) | 1 | 0 | 0
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 6 | 5 | 1
LOCALISED OEDEMA (General disorders) | 1 | 0 | 0
OEDEMA PERIPHERAL (General disorders) | 1 | 1 | 0
PAIN (General disorders) | 1 | 0 | 0
PYREXIA (General disorders) | 2 | 1 | 1
JAUNDICE (Hepatobiliary disorders) | 1 | 0 | 0
INFECTION (Infections and infestations) | 0 | 1 | 0
PERITONITIS BACTERIAL (Infections and infestations) | 0 | 1 | 0
PNEUMONIA (Infections and infestations) | 3 | 0 | 1
SEPSIS (Infections and infestations) | 0 | 0 | 1
SUPERINFECTION (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 1 | 0 | 0
BONE CONTUSION (Injury, poisoning and procedural complications) | 0 | 0 | 1
JAW FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 | 0 | 0
WEIGHT DECREASED (Investigations) | 0 | 1 | 0
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 | 1 | 1
DEHYDRATION (Metabolism and nutrition disorders) | 1 | 1 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0
HYPOVOLAEMIA (Metabolism and nutrition disorders) | 0 | 1 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
ALVEOLAR SOFT PART SARCOMA METASTATIC (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
TUMOUR HAEMORRHAGE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
COGNITIVE DISORDER (Nervous system disorders) | 0 | 1 | 0
SCIATICA (Nervous system disorders) | 0 | 0 | 1
DELIRIUM (Psychiatric disorders) | 0 | 1 | 0
DISORIENTATION (Psychiatric disorders) | 0 | 1 | 0
FEAR (Psychiatric disorders) | 1 | 0 | 0
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 2 | 0 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
CAPILLARY LEAK SYNDROME (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (N=37) | Arm II (N=24) | Arm III (N=10)
ANAEMIA (Blood and lymphatic system disorders) | 8 | 9 | 3
ANAEMIA OF MALIGNANT DISEASE (Blood and lymphatic system disorders) | 1 | 2 | 0
LEUKOPENIA (Blood and lymphatic system disorders) | 3 | 1 | 1
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 | 2 | 0
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 5 | 0 | 0
BUNDLE BRANCH BLOCK RIGHT (Cardiac disorders) | 0 | 0 | 1
CARDIOMEGALY (Cardiac disorders) | 0 | 0 | 1
SINUS BRADYCARDIA (Cardiac disorders) | 0 | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 1 | 0 | 2
CUSHING'S SYNDROME (Endocrine disorders) | 0 | 0 | 1
HYPERTHYROIDISM (Endocrine disorders) | 1 | 1 | 1
TOXIC NODULAR GOITRE (Endocrine disorders) | 0 | 0 | 1
LACRIMATION INCREASED (Eye disorders) | 0 | 0 | 1
MYOPIA (Eye disorders) | 0 | 0 | 1
VISION BLURRED (Eye disorders) | 0 | 0 | 1
VISUAL IMPAIRMENT (Eye disorders) | 0 | 0 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 4 | 7 | 3
APHTHOUS ULCER (Gastrointestinal disorders) | 3 | 0 | 1
ASCITES (Gastrointestinal disorders) | 1 | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 1 | 3 | 2
DIARRHOEA (Gastrointestinal disorders) | 5 | 6 | 3
DRY MOUTH (Gastrointestinal disorders) | 1 | 3 | 1
DYSPEPSIA (Gastrointestinal disorders) | 0 | 1 | 1
DYSPHAGIA (Gastrointestinal disorders) | 2 | 0 | 1
FLATULENCE (Gastrointestinal disorders) | 1 | 3 | 0
GASTROINTESTINAL DISORDER (Gastrointestinal disorders) | 0 | 0 | 1
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 | 0 | 1
MOUTH ULCERATION (Gastrointestinal disorders) | 0 | 0 | 1
NAUSEA (Gastrointestinal disorders) | 8 | 8 | 3
PROCTITIS (Gastrointestinal disorders) | 0 | 0 | 1
STOMATITIS (Gastrointestinal disorders) | 10 | 4 | 5
TOOTHACHE (Gastrointestinal disorders) | 2 | 0 | 0
VOMITING (Gastrointestinal disorders) | 6 | 5 | 3
ASTHENIA (General disorders) | 3 | 1 | 1
CHEST PAIN (General disorders) | 0 | 0 | 2
CHILLS (General disorders) | 1 | 1 | 1
DYSPLASIA (General disorders) | 0 | 0 | 1
FATIGUE (General disorders) | 10 | 9 | 5
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 3 | 1 | 0
GENERALISED OEDEMA (General disorders) | 2 | 0 | 0
IMPAIRED HEALING (General disorders) | 0 | 0 | 1
MEDICAL DEVICE PAIN (General disorders) | 0 | 0 | 1
MUCOSAL INFLAMMATION (General disorders) | 10 | 4 | 3
NON-CARDIAC CHEST PAIN (General disorders) | 1 | 0 | 1
OEDEMA PERIPHERAL (General disorders) | 6 | 6 | 3
PAIN (General disorders) | 3 | 0 | 1
PERIPHERAL SWELLING (General disorders) | 1 | 0 | 1
PYREXIA (General disorders) | 10 | 3 | 3
HEPATIC LESION (Hepatobiliary disorders) | 0 | 0 | 1
CONTRAST MEDIA ALLERGY (Immune system disorders) | 0 | 1 | 2
BRONCHITIS (Infections and infestations) | 4 | 1 | 0
CHRONIC SINUSITIS (Infections and infestations) | 0 | 0 | 1
CYSTITIS (Infections and infestations) | 1 | 1 | 2
FEBRILE INFECTION (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS (Infections and infestations) | 0 | 0 | 1
GASTROENTERITIS VIRAL (Infections and infestations) | 0 | 0 | 1
INFLUENZA (Infections and infestations) | 0 | 0 | 1
ORAL INFECTION (Infections and infestations) | 0 | 0 | 1
PHARYNGITIS (Infections and infestations) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 1 | 0 | 2
RHINITIS (Infections and infestations) | 1 | 0 | 1
SINUSITIS (Infections and infestations) | 0 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 3 | 0 | 1
VIRAL UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 1 | 5
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 0 | 0 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 0 | 0
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 4 | 0 | 1
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 3 | 3 | 0
BLOOD CHOLESTEROL INCREASED (Investigations) | 1 | 0 | 1
BLOOD CREATININE INCREASED (Investigations) | 3 | 1 | 0
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 4 | 3 | 0
C-REACTIVE PROTEIN INCREASED (Investigations) | 4 | 7 | 1
CLOSTRIDIUM TEST POSITIVE (Investigations) | 0 | 0 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 6 | 3 | 0
TRANSAMINASES INCREASED (Investigations) | 5 | 5 | 2
WEIGHT DECREASED (Investigations) | 7 | 7 | 1
CACHEXIA (Metabolism and nutrition disorders) | 0 | 2 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 13 | 6 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 | 0 | 0
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 | 2 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 10 | 5 | 0
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 0 | 1
TYPE 1 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 | 0 | 1
MUSCULOSKELETAL DISORDER (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 2 | 0 | 3
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
METASTASES TO CENTRAL NERVOUS SYSTEM (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
TUMOUR PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
DYSAESTHESIA (Nervous system disorders) | 1 | 0 | 1
DYSGEUSIA (Nervous system disorders) | 3 | 4 | 1
HEADACHE (Nervous system disorders) | 4 | 2 | 5
MIGRAINE (Nervous system disorders) | 0 | 1 | 1
SEIZURE (Nervous system disorders) | 0 | 0 | 1
DEPRESSION (Psychiatric disorders) | 1 | 1 | 1
INSOMNIA (Psychiatric disorders) | 0 | 0 | 1
SLEEP DISORDER (Psychiatric disorders) | 2 | 2 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 1 | 2 | 0
DYSURIA (Renal and urinary disorders) | 1 | 1 | 1
NOCTURIA (Renal and urinary disorders) | 3 | 3 | 0
URINARY RETENTION (Renal and urinary disorders) | 0 | 2 | 0
AMENORRHOEA (Reproductive system and breast disorders) | 0 | 0 | 1
MENORRHAGIA (Reproductive system and breast disorders) | 0 | 0 | 1
VAGINAL DISCHARGE (Reproductive system and breast disorders) | 0 | 0 | 1
VULVOVAGINAL INFLAMMATION (Reproductive system and breast disorders) | 0 | 0 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 5
DRY THROAT (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 2
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 1
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
PLEURISY (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
ACNE (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
DRY SKIN (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
ECZEMA (Skin and subcutaneous tissue disorders) | 3 | 0 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 2 | 0
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
PRURITUS (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
RASH (Skin and subcutaneous tissue disorders) | 8 | 5 | 3
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 0 | 0 | 1
HAEMATOMA (Vascular disorders) | 0 | 0 | 1
LYMPHOEDEMA (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2013-08-27): https://cdn.clinicaltrials.gov/large-docs/19/NCT00767819/Prot_000.pdf
  • Statistical Analysis Plan (2011-07-07): https://cdn.clinicaltrials.gov/large-docs/19/NCT00767819/SAP_001.pdf